CLINICAL TRIAL: NCT07005531
Title: Impact of Ultrasound-Guided Microbubble Clearance During CRRT Circuit Priming on Filter Lifespan: A Randomized Crossover Pilot Trial
Brief Title: Ultrasound-Guided Microbubble Removal and Filter Lifespan During CRRT: A Pilot Crossover Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Wannan Medical College (Other)
Responsible Party: Principal Investigator, Qiancheng Xu, Principal Investigator, First Affiliated Hospital of Wannan Medical College
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 202581
Record Dates: First submitted 2025-05-18; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Acute Kidney Injury; Continuous Renal Replacement Therapy (CRRT); Filter Clotting; Microbubbles; Ultrasound-Guided Microbubble Removal
Keywords: Continuous Renal Replacement Therapy (CRRT); Filter Lifespan; Microbubbles; Ultrasound Guidance; Filter Clotting; Circuit Priming; Critical Care; Randomized Crossover Trial
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Priming Group (No Intervention): CRRT circuits are primed using the standard visual inspection and manual bubble removal method without ultrasound guidance.
- Ultrasound-Guided Microbubble Removal Group (Experimental): CRRT circuits are primed with real-time ultrasound monitoring to detect and guide the removal of residual microbubbles before treatment.
  Interventions: Procedure: Ultrasound-Guided Microbubble Clearance During Circuit Priming

INTERVENTIONS:
Procedure: Ultrasound-Guided Microbubble Clearance During Circuit Priming — CRRT circuits will be primed under real-time ultrasound monitoring. A portable ultrasound probe will be used to scan key points in the circuit and filter to detect and guide the removal of residual microbubbles before treatment. The process is considered complete when three consecutive scans (at 2-minute intervals) show no detectable microbubbles.
  Arms: Ultrasound-Guided Microbubble Removal Group

SUMMARY:
What is this study about? This study is designed to evaluate whether ultrasound-guided removal of microbubbles during circuit priming in Continuous Renal Replacement Therapy (CRRT) can extend the filter lifespan for critically ill patients who require CRRT. The investigators aim to determine if this technique improves the duration of effective filter use and reduces complications related to filter clotting.

Who can join? Adults (18 years or older) admitted to the Intensive Care Unit (ICU) and diagnosed with acute kidney injury (AKI) or chronic kidney failure (CKD) who require CRRT and are expected to undergo at least two sessions of CRRT treatment.

Participants or their legal representatives must provide signed informed consent.

Who cannot join? Patients with severe coagulation disorders, platelet count <30×10^9/L, contraindications to anticoagulation, significant changes in clinical scores or blood tests between CRRT sessions, or any other condition deemed unsuitable by the investigator.

What will happen during the study?

Two Treatment Methods:

Conventional Priming (Control): The CRRT circuit will be primed following the standard visual bubble inspection protocol.

Ultrasound-Guided Priming (Intervention): The circuit will be primed using real-time ultrasound to detect and remove microbubbles from key locations.

Each participant will receive both interventions in random order, separated by a washout period of at least 24 hours.

Safe and Routine Monitoring:

Ultrasound scans will be performed on the filter and circuit to guide microbubble removal.

Standardized CRRT treatment protocols, including filter type and anticoagulation regimen, will be used for all sessions.

Other Data Collection:

Patient information (e.g., age, sex, medical history, APACHE II score) CRRT treatment details (e.g., filter lifespan, filter clotting incidence, coagulation parameters) Monitoring of adverse events and clinical outcomes (including 28-day survival and treatment costs) What are the benefits and risks? Benefits: This study may provide evidence for a simple, non-invasive method to reduce filter clotting, improve CRRT efficiency, and enhance patient outcomes.

Risks: Ultrasound monitoring is non-invasive and does not add risk beyond standard care. All procedures are standard clinical practice.

Your Rights and Safety Voluntary Participation: Participation is voluntary; withdrawal is allowed at any time without affecting clinical care.

Ethical Approval: The study protocol is reviewed and approved by the hospital's ethics committee.

Confidentiality: All personal information and test results will be kept confidential.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, regardless of sex;
* Admission to the intensive care unit (ICU) with a diagnosis of acute kidney injury (AKI) or chronic kidney disease (CKD) requiring continuous renal replacement therapy (CRRT);
* Expected to receive at least two sessions of CRRT;
* Written informed consent obtained from the patient or their legally authorized representative.

Exclusion Criteria:

* Presence of severe coagulopathy (such as disseminated intravascular coagulation, DIC) or platelet count <30×10^9/L;
* Contraindications to anticoagulation therapy;
* Change in APACHE II score >5 points, or changes in coagulation parameters and platelet count exceeding 20% between the two treatment sessions;
* Any other condition deemed unsuitable for participation by the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2026-06-29 (Estimated); Study Completion 2026-06-29 (Estimated)

PRIMARY OUTCOMES:
Filter Lifespan | For each CRRT session, up to a maximum of 72 hours per session.
  Time (in hours) from the start of CRRT treatment to filter failure (defined as filter clotting requiring replacement, or completion of prescribed treatment).
Feasibility of Ultrasound-Guided Microbubble Clearance | Peri-procedural (from initiation to completion of each CRRT session)
  Feasibility will be evaluated by the proportion of CRRT sessions in which microbubble clearance is completed according to predefined ultrasound scanning criteria (three consecutive scans at 10-minute intervals without detectable microbubbles). Assessment is based on procedure documentation and saved ultrasound images.

SECONDARY OUTCOMES:
Incidence of Filter Clotting | For each CRRT session, up to a maximum of 72 hours per session.
  Number and proportion of CRRT circuits with filter clotting events requiring early replacement.
28-Day Survival Rate | Day 28 after enrollment.
  Proportion of patients surviving at 28 days after enrollment.

IPD SHARING:
Plan to Share IPD: No